CLINICAL TRIAL: NCT00314353
Title: Randomized Phase II Clinical Trial of Bevacizumab Combined With Capecitabine and Either Oxaliplatin or Irinotecan as First Line Treatment for Metastatic Colorectal Cancer
Brief Title: Study of Bevacizumab Combined With Capecitabine and Either Oxaliplatin or Irinotecan as First Course of Treatment for Patients With Colorectal Cancer That Has Spread Beyond the Colon
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed early due to low enrollment and new information regarding the benefit of the study regimen.
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Genentech, Inc. (Industry); Hoffmann-La Roche (Industry); International Drug Development Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FC-BV-003
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2008-12-02 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Neoplasms
Keywords: NSABP; bevacizumab; capecitabine; oxaliplatin; irinotecan; rectal cancer; colon cancer; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine
- 2 (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Irinotecan

INTERVENTIONS:
Drug: Bevacizumab — 7.5 mg/kg IV Day 1 every 21 days for eight cycles*
  *For patients with stable or responding disease after 8 cycles, continue bevacizumab at the same dose levels until disease progression.
  Other Names: Avastin
Drug: Oxaliplatin — 130 mg/m2 IV Day 1 every 21 days for eight cycles
  Other Names: Eloxatin
  Arms: 1
Drug: Capecitabine — 850 mg/m2 po BID Days 1-14 every 21 days for eight cycles*#
  *For patients with stable or responding disease after 8 cycles, continue capecitabine at the same dose levels until disease progression.
  #For patients with baseline calculated creatinine clearance of 30-50 mL/min, the starting dose will be reduced to 650 mg/m2 BID
  Other Names: Xeloda
Drug: Irinotecan — 200 mg/m2 IV Day 1 every 21 days for eight cycles
  Other Names: Camptosar
  Arms: 2

SUMMARY:
Bevacizumab is an angiogenesis inhibitor which means it works to stop blood vessel formation in tumors. Without new blood vessels, the growth of a tumor is slowed. Chemotherapy works to kill cancer cells directly. This study is being done to see how colorectal cancer responds to treatment with the combination of bevacizumab and chemotherapy.

DETAILED DESCRIPTION:
Due to greater patient convenience and favorable toxicity profiles, clinical practice has seen an increased use of the combinations of capecitabine with oxaliplatin (CAPOX) and capecitabine with irinotecan (CAPIRI). Given the data documenting the improved efficacy for 5-FU based chemotherapy in combination with bevacizumab, it is important to investigate the potential advantages of adding this agent to regimens containing capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of colon or rectal cancer from either the colon or rectum or a metastatic site (beyond the colon or rectum)
* Evidence of adequate organ function (such as liver, kidneys, etc.)

Exclusion Criteria:

* Diagnosis of anal cancer
* Patients who are candidates for surgery
* Patients who have received previous treatments
* Pregnant or lactating women
* History of chronic disease(s) or other serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (1):
- NSABP Operations Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Protocol Therapy (8 Cycles)
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Started | 4 | 3
Completed | 2 (COMPLETED refers to the participants completing 8 cycles of therapy.) | 0 (COMPLETED refers to the participants completing 8 cycles of therapy.)
Not Completed | 2 | 3
Period: Follow-up
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Started | 3 (2 participants who completed 8 cycles plus 1 participant who did not complete 8 cycles therapy.) | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.0) | 63.0 (13.2) | 64.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: One-year Progression-free Survival (PFS)
Description: Outcome measure was not assessed due to early study closure. The study was closed early due to low enrollment and new information regarding the benefit of the study regimen.
Time Frame: Unevaluable - accrual ended early due to slow accrual rate and before accrual goal was met.
Population: Primary outcome measure was not assessed due to early study closure. The study was closed early due to low enrollment and new information regarding the benefit of the study regimen.
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Objective Response Rate
Time Frame: Unevaluable - accrual ended early due to slow accrual rate and before accrual goal was met.
Population: Outcome measure was not assessed due to early study closure. The study was closed early due to low enrollment and new information regarding the benefit of the study regimen.
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Toxicity - Adverse Events
Time Frame: Assessments before each cycle of chemotherapy, after every third dose of bevacizumab (if given alone), and final adverse event assessment 3 months after the last dose of bevacizumab
Population: as for outcome 2
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Time Frame: Unevaluable - accrual ended early due to slow accrual rate and before accrual goal was met.
Population: as for outcome 2
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response
Time Frame: Unevaluable - accrual ended early due to slow accrual rate and before accrual goal was met.
Population: as for outcome 2
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not assessed due to early study closure. The study was closed early due to low enrollment and new information regarding the benefit of the study regimen.
Arm/Group | Capecitabine, Oxaliplatin, Bevacizumab | Capecitabine, Irinotecan, Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was closed early due to low enrollment and new information regarding the benefit of the study regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less